CLINICAL TRIAL: NCT04135612
Title: The Use of Smartphone Based Communication for Encouragement of Breastfeeding and Early Detection of Post-partum Depression- A Randomized Control Trial
Brief Title: The Impact of a Daily Smartphone-based Communication Among Postpartum Women on Breastfeeding Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0026-19-WOMC
Record Dates: First submitted 2019-09-01; First posted 2019-10-22 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Breast Feeding, Exclusive; Post Partum Depression
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone group (Experimental): application installed to their smartphones. This application will be in Hebrew language, simple to use, and specifically designed to the needs of the current study.
  Each patient will document each evening her lactation performance during the day, and the App will generate a daily report transmitted by email every evening to our computerized research database. Every evening the patient will receive via email an individualized feedback from our team regarding her lactation. This feedback could include: reassurance and positive feedback and lactation tips in attempt to optimize specific obstacles. In addition, patients will be encouraged to use the platform to ask questions and receive immediate answers regarding any aspect lactation. As per the study protocol, medical treatment will only be initiated in a formal clinic appointment and not via the application.
  Interventions: Other: Smartphone based communication
- Control group (No Intervention): The routine prenatal care provided by our institute includes lactation consulting during the 48-72 hour postpartum hospitalization.

INTERVENTIONS:
Other: Smartphone based communication — Each patient will document each evening her lactation performance during the day, and the App will generate a daily report transmitted by email every evening to our computerized research database. Every evening the patient will receive via email an individualized feedback from our team regarding her lactation. This feedback could include: reassurance and positive feedback and lactation tips in attempt to optimize specific obstacles.
  Arms: Smartphone group

SUMMARY:
We will aim to study the impact of introducing a smartphone-based daily feedback and communication platform between postpartum women delivering at our institute and a multidisciplinary breastfeeding-support team (obstetricians, neonatologists, midwives, lactation consultants, nurses, and psychologist) on breastfeeding rates.

DETAILED DESCRIPTION:
Our study will aim to introduce a smartphone-based daily feedback and communication platform between postpartum women delivering at our institute and a multidisciplinary breastfeeding-support team. This team will include: an obstetrician specialized in maternal-fetal medicine, a general obstetrician, two certified midwives, two certified lactation-consultants, a neonatologist, and a psychologist. Our vision and hypothesis for the current study- is that an intimate personalized daily communication and feedback platform between each woman and the support team will improve the rates of initiation of lactation and of full/partial lactation at various time points postpartum.

Geographic area - A university affiliated hospital in southern Tel-Aviv that serves a population of over 500,000 people. Our annual delivery volume is 5000 deliveries with a 22% CS rate. The population is heterogeneous and consists of a high rate of women with intermediate-low income as well as a population of refugees from Africa (mostly Eritrea), both populations still have a very high rate of smartphone owners based on our previous experience.

Methods- Prospective, single-center randomized controlled trial. Eligibility will be limited to women expressing wish to breastfeed, with singleton gestations, delivering > 37 weeks with no other maternal/neonatal significant morbidities.

Study design and group assignment -Women meeting inclusion criteria who own a smartphone will be approached for recruitment on postpartum day 1. After obtaining a written informed consent, patients will be randomly assigned either to the intervention group (smartphone group) or to the control group in a 1:1 ratio. A blocked randomization scheme will be created using a computer-generated list of random numbers.

The routine prenatal care provided by our institute includes lactation consulting during the 48-72 hour postpartum hospitalization. Patients allocated to the control group will receive the aforementioned care. Patients assigned to the smartphone group will receive our standard care, and in addition will have an application installed to their smartphones. This application will be in Hebrew language, simple to use, and specifically designed to the needs of the current study.

All patients will receive a demonstration regarding the use of the application from one of our research coordinators, in addition to a detailed information brochure.

the patient will receive via email an individualized feedback from our team regarding her lactation. This feedback could include: reassurance and positive feedback and lactation tips in attempt to optimize specific obstacles. In addition, patients will be encouraged to use the platform to ask questions and receive immediate answers regarding any aspect lactation.

Primary outcome- Lactation at 3 months postpartum Secondary outcomes Full/partial lactation at 2 weeks, 4 weeks, 6 weeks, 3 months, and 6 months and a variety of outcomes regarding neonatal health, maternal health, emotional status and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* women expressing wish to breastfeed, with singleton gestations, delivering > 37 weeks with no other maternal/neonatal significant morbidities.

Exclusion Criteria:

* refusal to participate
* no smartphone availability

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 224 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
breastfeeding rates | 3 months
  Full or partial breastfeeding at fixed intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson medical center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miremberg H, Yirmiya K, Rona S, Gonen N, Marom O, Pohol A, Kovo M, Bar J, Weiner E. Smartphone-based counseling and support platform and the effect on postpartum lactation: a randomized controlled trial. Am J Obstet Gynecol MFM. 2022 Mar;4(2):100543. doi: 10.1016/j.ajogmf.2021.100543. Epub 2021 Dec 4. PMID 34871782